CLINICAL TRIAL: NCT01481831
Title: A Multi-center, Stratified Randomized, Controlled Study to Evaluate the Efficacy and Safety of Palonosetron Hydrochloride in the Prevention of Nausea and Vomiting Associated With Moderate and Highly Emetogenic Chemotherapy in China
Brief Title: Efficacy and Safety of Palonosetron Hydrochloride in the Prevention of Nausea and Vomiting
Acronym: ESPNV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: JiangSu Chia-Tai Tianqin Pharmacy Co.Ltd (Unknown)
Responsible Party: Principal Investigator, Zhan Wang, Principal Investigator, Shanghai Changzheng Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: zhiruo
Record Dates: First submitted 2011-10-28; First posted 2011-11-30 (Estimated); Last update posted 2012-12-31 (Estimated); Status verified 2012-12

CONDITIONS: Neoplasms; Chemotherapy-Induced Nausea and Vomiting
MeSH Terms: conditions — Neoplasms; Vomiting | interventions — Palonosetron

ARMS (4):
- H PALO day 1 (Active Comparator): Highly Emetogenic Arm, Palonosetron 0.25mg IV*1 dose on day 1
  Interventions: Drug: Palonosetron Hydrochloride
- H PALO day 1,3,5 (Experimental): Highly Emetogenic Arm, Palonosetron 0.25mg IV*3 doses on days 1,3 and 5
  Interventions: Drug: Palonosetron Hydrochloride
- M PALO day 1 (Active Comparator): Moderately Emetogenic Arm, Palonosetron 0.25mg IV*1 dose on day 1
  Interventions: Drug: Palonosetron Hydrochloride
- M PALO day 1,3,5 (Experimental): Moderately Emetogenic Arm, Palonosetron 0.25mg IV*3 doses on days 1,3 and 5
  Interventions: Drug: Palonosetron Hydrochloride

INTERVENTIONS:
Drug: Palonosetron Hydrochloride — 0.25 mg IV*1 dose on day 1, 30 minutes prior to the administration of the major chemotherapeutic agent.
  Arms: H PALO day 1; M PALO day 1
Drug: Palonosetron Hydrochloride — 0.25mg IV*3 doses on days 1,3 and 5,30 minutes prior to the administration of the major chemotherapeutic agent.
  Arms: H PALO day 1,3,5; M PALO day 1,3,5

SUMMARY:
This purpose of this study is to evaluate the efficacy and safety of single and repeated doses of palonosetron hydrochloride in preventing nausea and vomiting caused by moderate and highly emetogenic chemotherapy in patients.

DETAILED DESCRIPTION:
Group I (Highly Emetogenic Chemotherapy): Patients that accepted chemotherapy including Cisplatin≥50mg/m2, Carmustine>250mg/m2, Cyclophosphamide>1500mg/m2, Dacarbazine>60mg/m2, Doxorubicin>60mg/m2, Epirubicin>90mg/m2, IFO≥10g/m2 or AC program.

Group II (Moderately Emetogenic Chemotherapy): Patients that accepted chemotherapy including any dose of Carboplatin, Daunorubicin, Oaliplatin, Irinotecan, or Doxorubicin<60mg/m2(not include liposomal doxorubicin), Epirubicin≤90mg/m2, Carmustine≤250mg/m2, Methotrexate≥250mg/m2, Cyclophosphamide≤1500mg/m2, Arabinoside>200mg/m2, IFO<10g/m2, Cisplatin≥50mg/m2.

Total subjects: 1000, single dose of palonosetron group of 500 patients, repeated doses of palonosetron group of 500 patients. According to the study subjects receiving highly emetogenic chemotherapy or moderately emetogenic chemotherapy, subjects are stratified randomize.

ELIGIBILITY:
Inclusion Criteria:

1. Patients candidates to a chemotherapy treatment, with histologically or cytologically confirmed malignant disease;
2. The concrete chemotherapy plan does not limited, group I (Highly Emetogenic Chemotherapy), group II (Moderately Emetogenic Chemotherapy);
3. Male or female aged 18-75 years, ECOG≤2, estimates survival time≥3 months;
4. WBC≥3.0×109/L, ANC≥1.5×109/L, PLT≥80×109/L, total bilirubin≤1.5×ULN(Normal value upper limit), AST and ALT≤2.5×ULN(With transferability liver cancer≤5×ULN), Cr and BUN≤1.5×ULN, electrolyte and electrocardiogram are normal, conforms to the chemotherapy adaptation;
5. Patients have been apart from the previous chemotherapy to finish above 2 weeks (including 2 weeks);
6. Patients that voluntarily sign the consent form.

Exclusion Criteria:

1. Pregnancy, or patients during breast feeding;
2. Patients have accepted any radiotherapy during the experimental period;
3. Gastric outlet or intestinal obstruction;
4. Patients have serious heart diseases, liver kidney diseases, or metabolism function disorder;
5. Patients have epilepsy, or have been used psychotropic drug and calm drug;
6. Received any drugs with potential anti-emetic efficacy, or experienced any vomiting, nausea or retching in the 24 hours prior to chemotherapy;
7. Patients with transferability brain tumor, have vomiting caused by skull high pressure, or can not speak sickness situation and adverse reactions by self;
8. Patients have known hypersensitivity to 5-HT3 antagonists;
9. Patients have chemotherapy contraindications;
10. Patients are participating, or have participated in other Clinical studies of new drugs within 2 weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 599 (Actual)
Dates: Start 2011-07; Primary Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Complete Response rate | 2-7 days
  defined as no emetic episode and no use of rescue medication

SECONDARY OUTCOMES:
Complete Response rate | 0-24 hours, 0-7 days
  defined as no emetic episode and no use of rescue medication

CONTACTS AND LOCATIONS:
Locations (18):
- China (18):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Chinese Academy of Medical Sciences Cancer Hospital, Beijing, Beijing Municipality
  - Chinese PLA 301 Hospital, Beijing, Beijing Municipality
  - Chinese PLA 307 Hospital, Beijing, Beijing Municipality
  - Chinese PLA Navy General Hospital, Beijing, Beijing Municipality
  - Fuzhou General Hospital of Nanjing Military Command, Fuzhou, Fujian
  - Guangxi Cancer Hospital, Nanning, Guangxi
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Nanjing General Hospital of Nanjing Military Command, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Fourth People's Hospital of Wuxi, Wuxi, Jiangsu
  - Shandong Cancer Hospital, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - The Affiliated Hospital of Medical College Qingdao University, Qingdao, Shandong
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - Shanghai Xinhua Hospital, Shanghai, Shanghai Municipality
  - Tangdu Hospital of Fourth Military Medical University, Xian, Shanxi